CLINICAL TRIAL: NCT04606316
Title: A Phase Ib Clinical Trial to Evaluate Early Immunologic Pharmacodynamic Parameters Following Neoadjuvant Anti-PD-1 (Nivolumab), or the Combination of Anti-PD-1 Plus Anti-CTLA-4 (Nivolumab Plus Ipilimumab) in Patients With Surgically Accessible Glioblastoma
Brief Title: Surgical Nivolumab And Ipilimumab For Recurrent GBM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Patrick Wen, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Patrick Wen, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-494
Record Dates: First submitted 2020-10-24; First posted 2020-10-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; GBM; Glioblastoma Multiforme; Grade IV Astrocytoma
Keywords: Glioblastoma; GBM; Glioblastoma Multiforme; Grade IV Astrocytoma
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab; Ipilimumab; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The neoadjuvant treatment administered prior to surgery will be blinded. The participants, Sponsor, site investigators, and site staff will not know the treatment administered. An assigned Site Investigational Pharmacist will not be blinded. Designated staff of the DF/HCC Office of Data Quality will be unblinded to facilitate randomization and safety monitoring. Treatment after surgery is not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nivolumab and Ipilimumab Before and After Surgery (Experimental): One dose of nivolumab plus ipilimumab will be administered 14(±5) days before surgery.
  After surgery, participants receive nivolumab in combination with ipilimumab every 3 weeks for 9 weeks and then nivolumab alone every 4 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Procedure: Surgery
- Nivolumab and Placebo-Ipilimumab Before Surgery, Nivolumab After Surgery (Experimental): One dose of nivolumab plus placebo-ipilimumab will be administered 14(±5) days before surgery.
  After surgery, participants receive nivolumab in combination with ipilimumab every 3 weeks for 9 weeks and then nivolumab alone every 4 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab-Placebo; Procedure: Surgery
- Placebo-Nivolumab and Placebo-Ipilimumab Before Surgery, Nivolumab and Ipilimumab After Surgery (Experimental): One dose of placebo-nivolumab plus placebo-ipilimumab will be administered 14(±5) days before surgery.
  After surgery, participants receive nivolumab in combination with ipilimumab every 3 weeks for 9 weeks and then nivolumab alone every 4 weeks
  Interventions: Drug: Nivolumab-Placebo; Drug: Nivolumab; Drug: Ipilimumab-Placebo; Drug: Ipilimumab; Procedure: Surgery

INTERVENTIONS:
Drug: Nivolumab-Placebo — Intravenous (IV) solution that has no therapeutic effect, used as a control in testing investigational drug. One dose is received prior to surgery.
  Arms: Placebo-Nivolumab and Placebo-Ipilimumab Before Surgery, Nivolumab and Ipilimumab After Surgery
Drug: Nivolumab — Given as intravenous (IV) infusion into a vein.
  Other Names: Opdivo
Drug: Ipilimumab-Placebo — Intravenous (IV) solution that has no therapeutic effect, used as a control in testing investigational drug. One dose is received prior to surgery.
  Arms: Nivolumab and Placebo-Ipilimumab Before Surgery, Nivolumab After Surgery; Placebo-Nivolumab and Placebo-Ipilimumab Before Surgery, Nivolumab and Ipilimumab After Surgery
Drug: Ipilimumab — Given as intravenous (IV) infusion into a vein.
  Other Names: Yervoy
  Arms: Nivolumab and Ipilimumab Before and After Surgery; Placebo-Nivolumab and Placebo-Ipilimumab Before Surgery, Nivolumab and Ipilimumab After Surgery
Procedure: Surgery — Treatment of disease or injury by cutting, abrading, suturing, or otherwise physically changing body tissues and organs.
  Other Names: Resection

SUMMARY:
This research trial is studying the safety and effectiveness of nivolumab in combination with ipilimumab and surgery when used in the treatment of recurrent glioblastoma.

The names of the study drugs involved in this study are:

* Nivolumab
* Ipilimumab
* Placebo (IV solution with no medicine)
* Zr-89 Crefmirlimab berdoxam (optional sub-study)

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. It is expected that about 60 people will take part in this research study.

There are 3 study groups participating in this study and each group receives different study drugs. After screening, participants will be randomized into one of three study groups.

Participants will receive one of the following study treatments prior to undergoing surgery for tumor removal:

* Group A receives nivolumab plus ipilimumab
* Group B receives nivolumab plus placebo-ipilimumab
* Group C receives two placebo infusions, placebo-nivolumab plus placebo-ipilimumab

Neither the participant nor the research doctor will know which study drugs the participant will receive prior to surgery.

After recovering from surgery, participants will receive the following doses of study medication:

-- Nivolumab plus ipilimumab every 3 weeks for 3 doses followed by nivolumab every 4 weeks

This research study is a Phase Ib clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved the use of nivolumab or ipilimumab for your specific disease, but it has been approved for other uses.

Both nivolumab and ipilimumab are antibodies (types of human protein) that work to stop tumor cells from growing and multiplying by immunotherapy.

Immunotherapy is trying to have the body's own immune system work against tumor cells. Nivolumab and ipilimumab have been used in other research studies, and information from those other research studies suggest these drugs may help to stop glioblastoma cells from growing.

Subjects also have the option of undergoing Zr-89 Crefmirlimab berdoxam PET scans. This consists of one infusion with Zr-89 Crefmirlimab berdoxam followed by a PET scan prior to starting study treatment and another infusion with PET scan about 3 days prior to surgery.

The U.S. Food and Drug Administration (FDA) has not approved Zr-89 Crefmirlimab berdoxam as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed World Health Organization Grade IV IDH wildtype glioblastoma or variants including gliosarcoma or IDH wildtype glioma with molecularly features of glioblastoma.
* Previous first line therapy with at least radiotherapy.
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers.
* Be at first or second relapse. Note: Relapse is defined as progression following initial therapy (i.e., radiation ± chemotherapy).
* Participants must have shown unequivocal evidence for tumor progression by MRI per RANO criteria.
* Participants must have confirmation of availability of sufficient tissue from prior surgery revealing glioblastoma or variants for submission following registration. The following amount of tissue is required:

  * 1 formalin-fixed paraffin-embedded (FFPE) tumor tissue block (preferred) OR
  * 10 FFPE unstained slides (5 μm thick)
* An interval of at least 12 weeks from the completion of radiation therapy to registration unless there is unequivocal histologic confirmation of tumor progression.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia (which is common after therapy with temozolomide).
* An interval of at least 4 weeks (to registration) between prior surgical resection or one week for stereotactic biopsy.
* From registration, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 4 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies (including vaccines). No washout period required from tumor treating fields (TTF).
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have a Karnofsky performance status (KPS) ≥ 70.
* MRI within 14 days prior of registration.
* All screening labs should be performed within 14 days of registration and demonstrate adequate organ function as defined below:

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Serum creatinine OR measured or calculated a creatinine clearance (GFR can be used in place of creatinine or CrCl) ≤1.5 X institutional upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (Creatinine clearance should be calculated per institutional standard.)
  * Serum total bilirubin ≤ 1.5 X institutional ULN OR direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X institutional ULN OR ≤ 5 X institutional ULN for subjects with Gilberts syndrome
  * Albumin ≥ 2.5 mg/dL
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment if she considered not of child bearing potential.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during study treatment and for 5 months after study discontinuation. Highly effective contraception is defined as either:

  * True Abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
  * Sterilization: Surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment (as described above).
  * Male Partner Sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that participant.
  * Use of a combination of any two of the following:

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
    * Appropriate hormonal contraceptives (including any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent - including oral, subcutaneous, intrauterine, or intramuscular agents).
* Male subjects should agree to use adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of therapy.

Exclusion Criteria:

* IDH mutation by immunohistochemistry.
* Current or planned participation in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency.
* Has tumor primarily localized to the brainstem or spinal cord.
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc.) within six months of registration.
* Has received bevacizumab or aflibercept. VEGFR inhibitors are allowed.
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent at the time of registration.
* Has received prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection or convection enhanced delivery.
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of registration.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of registration.
* Has a known additional malignancy that is progressing or requires active treatment. Those patients whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen will be eligible including, but not limited to, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized prostate cancer not requiring treatment, or in situ cervical cancer that has undergone potentially curative therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Examples include but are not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant, breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 5 months after the last dose of trial treatment. It is unknown whether nivolumab and/or ipilimumab is excreted in human milk or may have adverse effects on a fetus in utero. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant or fetus, these subjects are not eligible for enrollment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-Associated Antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to registration.
* Has a known hypersensitivity to any of the study therapy products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Infiltrating T Lymphocyte (TIL) Density | 24 Months
  TIL density will be assessed and compared between the three arms using the Two-sample t-Test.
Safety of Study Drug Therapy | 24 Months
  Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Safety will be assessed by quantifying the toxicities and grades experienced by participants who have received at least one dose of study treatment.

SECONDARY OUTCOMES:
Cell Cycle-Related Genetic Signature within the Tumor Microenvironment | 24 months
  Multiplex IHC staining will be performed on tumor tissue to evaluate the influence of the neoadjuvant administration on the cell cycle-related genetic signature within the tumor microenvironment of recurrent glioblastoma.
Percentage of Progression Free Survival (PFS-6) | 24 months
  PFS-6 will be assessed using pooled data in comparison to appropriate historical controls. Percent PFS-6 will be estimated and compared using the Exact Binomial Test.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu